CLINICAL TRIAL: NCT03510065
Title: Post Market Clinical Follow-Up Study Prevision®
Brief Title: Prevision® PMCF Study
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1508
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Survival, Prosthesis
Keywords: hip arthroplasty; revision arthroplasty; survival
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Prevision® — One time Evaluation with documentation of one follow-up visit

SUMMARY:
Monocentric, non-interventional Post-Market Clinical Follow-Up (PMCF) Study on past implantations of the Prevision® prosthesis; the survival rate of the Prevision® prosthesis shall be evaluated and compared to literature results on comparable Revision stems.

ELIGIBILITY:
Inclusion:

* Patient received a Prevision® Hip Stem (curved or straight) between 2002 an 2012
* Patient gave his written consent for study participation

Exclusion:

- none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving a Prevision® stem between 2002 and 2012
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Prevision® survival | 4-14 years after implantation
  Kaplan Meier Survival Rate, retrospective Analysis of Patients operated between 2002 and 2012

SECONDARY OUTCOMES:
Clinical Results | 4-14 years after implantation
  Harris Hip Score: The score covers pain, function, absence of deformity, and range of motion. Pain is measured as pain severity and its effect on activities and need for pain medication.
  Hip function score consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction.
  There are 10 items. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
Ectopic Ossification | 4-14 years after implantation
  Radiological Results, Ectopic Ossification acc. to Brooker; retrospective Analysis of Patients operated between 2002 and 2012
Sinking / Migration of the Stem | 4-14 years after implantation
  Radiological Results, Sinking / Migration of the Stem in [mm], Comparison to x-ray at Hospital discharge where available, retrospective Analysis of Patients operated between 2002 and 2012
Radiological Evaluation of the Stem | 4-14 years after implantation
  Radiological Results of Radiolucent Lines, Osteolysis, Hypertrophy, Decrease of corticalis thickness, Cyst; retrospective Analysis of Patients operated between 2002 and 2012
Quality of Life | 4-14 years after implantation
  Measured by EQ-5D-5L: The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Pain | 4-14 years after implantation
  Pain in the hip Joint, measured by Visual Analogue Scale: The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
Adverse Events | 4-14 years after implantation
  Documentation of any Adverse event
Serious Adverse Events | 4-14 years after implantation
  Documentation of any Serious Adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Bad Hersfeld, Bad Hersfeld, Germany